CLINICAL TRIAL: NCT00277355
Title: A Multi-Center, Double-Blind, Pilot Study of Minocycline in Huntington's Disease
Brief Title: Pilot Study of Minocycline in Huntington's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit Cudkowicz (Network)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Merit Cudkowicz, Principal Investigator, Huntington Study Group
Organization: Huntington Study Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FD-R-002588; DOMINO
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Huntington Disease
Keywords: Study of Minocycline in Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): Minocycline (3:1 randomization) 100 mg capsules taken by mouth twice daily, 200 mg per day total for 18 months treatment duration.
  Interventions: Drug: minocycline
- Matching placebo (Placebo Comparator): Sugar pill manufactured to mimic minocycline, 1 capsule taken by mouth twice daily for 18 months treatment duration.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: minocycline — Minocycline: Oral; minocycline 100 mg capsules administered twice a day with the morning and evening meal (~ 8 hours apart)
  Arms: Minocycline
Drug: Matching placebo — Matching placebo 1 capsule twice daily, 18 months treatment duration.
  Arms: Matching placebo

SUMMARY:
This study is being conducted to assess the impact of minocycline on the progression of symptoms of HD. The study will also assess whether it is reasonable to continue with further study of minocycline in HD. We will measure the effect of minocycline on HD by measuring the change in Huntington's disease symptoms.

DETAILED DESCRIPTION:
The DOMINO study is a randomized, double-blind, multi-center, futility study of minocycline in patients with HD. Subjects will be randomized (3:1) to one of the two study arms: (1) the group that receives active minocycline (100 mg po b.i.d.), and (2) the group that receives placebo. Subjects will be enrolled over an approximate six-month period and remain on blinded study drug for 18 months. The primary analysis will involve a comparison of the change over time in TFC between the minocycline group and a fixed value determined from historical control data. A placebo group will also be included to facilitate blinding and to permit a descriptive assessment of the validity of the assumed change over time in historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical features of HD and a confirmatory family history of HD; and/or genetically confirmed HD
* Independently walking and fully self-sufficient in activities of daily living (eating, dressing, bathing)
* Able to take medication (capsules) by mouth

Exclusion Criteria:

* History of known hypersensitivity or intolerability to minocycline or known allergy to any tetracycline
* History of vestibular disease
* Subjects with underlying hematologic, hepatic or renal disease
* History of systemic lupus erythematosus (SLE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit E. Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (12):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - University of Texas Medical Branch at Galveston, Galveston, Texas
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Huntington Study Group. Minocycline safety and tolerability in Huntington disease. Neurology. 2004 Aug 10;63(3):547-9. doi: 10.1212/01.wnl.0000133403.30559.ff. PMID 15304592
- See also: The Huntington Study Group (HSG) is a non-profit group of physicians and other health care providers from medical centers in the U.S., Canada, Europe and Australia, experienced in the care of Huntington patients and dedicated to clinical research of HD. — http://www.Huntington-Study-Group.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2006 and June 2007 , 134 patients were screened and 114 subjects were randomized at 12 Huntington Study Group clinical sites.
Pre-assignment Details: 20 subjects were excluded from group assignment after screening: 14 failed inclusion criteria and 6 withdrew consent. Minocycline 90 days prior to baseline and open-label during trial not permitted. Other tetracyclines, investigational drugs, lithium, digoxin, methoflurane anesthesia, theophylline and lupus-symptom causing drugs not permitted.
Groups:
- Minocycline 100 mg Twice Daily: Minocycline 100 mg/twice daily (minocycline to placebo 3:1 ratio randomization).
- Matching Placebo Twice Daily: Matching placebo twice daily (minocycline to placebo 3:1 ratio randomization).
Period: Overall Study
Arm/Group | Minocycline 100 mg Twice Daily | Matching Placebo Twice Daily
Started | 87 | 27
Completed | 73 | 22
Not Completed | 14 | 5
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 5 | 0
Not completed — Death | 3 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Matching Placebo Twice Daily: Matching placebo twice daily (minocycline to placebo 3:1 ratio randomization.
- Total: Total of all reporting groups
Arm/Group | Minocycline 100 mg Twice Daily | Matching Placebo Twice Daily | Total
Number analyzed (Participants) | 87 | 27 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 25 | 110
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 47.1 (10.3) | 47.8 (10.6) | 47.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 15 | 61
  Male | 41 | 12 | 53
Region of Enrollment [Number; unit: participants]
  United States | 80 | 25 | 105
  Canada | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 18 in the Total Functional Capacity (TFC) Scale [LOCF Imputation Method]
Description: Establish preliminary estimate of minocycline's impact on progression of HD (measured by the change in Total Functional Capacity (TFC) score of Unified Huntington's Disease Rating Scale [UHDRS] between baseline & Month 18), and to assess futility of further study of minocycline. TFC consists of five ordinally scaled items assessing a person's capacity with: 1. occupation 2. financial affairs 3. domestic responsibilities 4. activities of daily living and 5. independent living. Total score ranges from zero (worst) to 13 (best).
Time Frame: Baseline to 18 months
Population: The primary analyses were performed according to the intent to treat principle and included all randomized subjects. Two strategies were used to address missing data: 1. Last observation carried forward (LOCF) was used to impute missing values and 2. A secondary method of regression-based multiple imputation was also used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline 100 mg Twice Daily | Matching Placebo Twice Daily
Number analyzed (Participants) | 87 | 27
units on a scale | 1.55 (1.85) | 1.15 (1.70)

2. Secondary Outcome: Change From Baseline to Month 18 in the Total Functional Capacity (TFC) Scale [Regression Based Multiple Imputation Method]
Description: TFC consists of five ordinally scaled items assessing a person's capacity with: (1) occupation; (2) financial affairs; (3) domestic responsibilities; (4) activities of daily living; and (5) independent living. Total score ranges from zero (worst) to 13 (best). Regression based imputation was used to impute missing values.
Time Frame: Baseline to 18 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline 100 mg Twice Daily | Matching Placebo Twice Daily
Number analyzed (Participants) | 87 | 27
units on a scale | 1.71 (1.96) | 1.15 (1.70)

ADVERSE EVENTS:
Time Frame: Baseline to 18 months
Arm/Group | Minocycline 100 mg Twice Daily | Matching Placebo Twice Daily
Serious Adverse Events (participants affected / at risk) | 11/87 | 1/27
Other Adverse Events (participants affected / at risk) | 74/87 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline 100 mg Twice Daily (N=87) | Matching Placebo Twice Daily (N=27)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deyhdration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Agitated depression (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aborted pregnancy (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline 100 mg Twice Daily (N=87) | Matching Placebo Twice Daily (N=27)
Dysphagia (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 7 | 0
Irritability (General disorders) | 5 | 1
Bronchitis (Infections and infestations) | 0 | 2
Gatrointestional viral (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 3 | 2
Nasophyngitis (Infections and infestations) | 5 | 3
Tooth abscess (Infections and infestations) | 0 | 2
Back injury (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 2
Fall (Injury, poisoning and procedural complications) | 15 | 6
Joint sprain (Injury, poisoning and procedural complications) | 3 | 3
Skin laceration (Injury, poisoning and procedural complications) | 2 | 4
Weight decreased (Investigations) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Balance disorder (Nervous system disorders) | 9 | 2
Chorea (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 7 | 1
Depressed mood (Psychiatric disorders) | 6 | 1
Depression (Psychiatric disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 8 | 2
Libido decreased (Psychiatric disorders) | 0 | 2
Obsessive thoughts (Psychiatric disorders) | 5 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No